CLINICAL TRIAL: NCT02418624
Title: A Phase I Followed by a Randomized Phase II Trial of Two Cycles Carboplatin-Olaparib Followed by Olaparib Monotherapy Versus Capecitabine in BRCA-1 or -2 Mutated Her2 Negative Advanced Breast Cancer as First Line Treatment
Brief Title: Phase I of Carboplatin-Olaparib Followed by Olaparib Monotherapy in Advanced Cancer
Acronym: REVIVAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14REV; NL50610.031.14 (Other: Netherlands CCMO); 2013-005590-41 (EudraCT Number)
Record Dates: First submitted 2015-03-09; First posted 2015-04-16 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Advanced Cancer
Keywords: breast cancer 1, early onset (BRCA1); breast cancer 2, early onset (BRCA2); homologous recombination deficiency; carboplatin; olaparib
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — Carboplatin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): carboplatin, olaparib
  Interventions: Drug: carboplatin, olaparib

INTERVENTIONS:
Drug: carboplatin, olaparib — 2 cycles of carboplatin and olaparib combination therapy followed by olaparib monotherapy.

SUMMARY:
A phase I trial to determine the recommended phase two dose of the combination of carboplatin and olaparib.

DETAILED DESCRIPTION:
A 3+3 dose escalation trial of 2 cycles (21 days) carboplatin and olaparib combination therapy, followed by olaparib monotherapy until progression or unacceptable toxicity in patients with advanced cancer.

ELIGIBILITY:
Inclusion criteria:

1. Histological or cytological proof of advanced cancer pre-treated with maximally one line of systemic chemotherapy in the advanced setting and any line of hormonal therapy for advanced disease, and potentially benefitting from olaparib-carboplatin combination therapy (prior (neo-)adjuvant chemotherapy is accepted and does not count as one line, since administered in early stage disease);
2. Age ≥ 18 years;
3. Able and willing to give written informed consent;
4. WHO performance status of 0, 1 or 2;
5. Able and willing to undergo blood sampling for PK and PD analysis;
6. Life expectancy ≥ 3 months, allowing adequate follow up of toxicity evaluation and antitumor activity;
7. Evaluable disease according to RECIST 1.1 criteria;
8. Minimal acceptable safety laboratory values

   1. ANC of ≥ 1.5 x 10^9 /L
   2. Hemoglobin of at least 6.2 mM and no transfusions in the last 28 days.
   3. Platelet count of ≥ 100 x 10^9 /L
   4. Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN (or < 3 x ULN in case of known Gilbert syndrome), ASAT and ALAT 2.5 x ULN (or <5 x ULN in case of liver metastasis)
   5. Renal function as defined by serum creatinine ≤1.5 x ULN or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula);
9. Negative pregnancy test (urine/serum) for female patients with childbearing potential;

Exclusion criteria

1. Any treatment with investigational drugs within 28 days prior to receiving the first dose of investigational treatment; or 21 days for standard (neo-)adjuvant chemotherapy, hormonal and immunotherapy;
2. Patients who have received high dose alkylating agents, a PARP1 inhibitor or carboplatin pretreatment; unless no progression on carboplatin had been observed during earlier treatment and the last carboplatin administration had been longer than 6 months ago;
3. Any current treatment with drugs that induce or inhibit the CYP3A4 system : http://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm#inVivo or APPENDIX IX
4. Women who have a positive pregnancy test (urine/serum) and/or who are breast feeding;
5. Unreliable contraceptive methods. Women and men enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: oral, injected or implanted hormonal methods, intra-uterine devices or systems, condom or other barrier contraceptive measures, sterilization and true abstinence)
6. Radiotherapy within the last four weeks prior to receiving the first dose of investigational treatment; except 1x8 Gy for pain palliation then a seven days interval should be maintained;
7. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
8. Patients with known active hepatitis B or C;
9. Recent myocardial infarction (< six months) or unstable angina;
10. Symptomatic brain metastases. If adequately treated with resection and/or irradiation and patients are at least four weeks completely free of symptoms of these metastases and without medication related to these metastases patients could be eligible if all other in- and exclusion criteria are obeyed.
11. Known leptomeningeal metastases.
12. Patients with myelodysplastic syndrome or acute myeloid leukemia
13. Any medical condition not yet specified above that is considered to possibly, probably or definitely interfere with study procedures, including adequate follow-up and compliance and/or would jeopardize safe treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | per doselevel of 3 to 6 patients (when 3-6 patients have completed DLT period of 3 weeks)
  The dose level at which more than 1/6 patients develop a dose limiting toxicity

SECONDARY OUTCOMES:
Pharmacokinetics (area under time-concentration curve (AUC)) | 1 year
  Pharmacokinetics (PK) measurements of olaparib alone and olaparib in combination with carboplatin
Pharmacodynamics (PAR (Poly(ADP) ribose) activation measured with the PAR assay) | 1 year
  PAR (Poly(ADP) ribose) activation measured with the PAR assay
Objective Response Rate | 1 year
  Objective Response Rate according to Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Linn, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] Schouten PC, Dackus GM, Marchetti S, van Tinteren H, Sonke GS, Schellens JH, Linn SC. A phase I followed by a randomized phase II trial of two cycles carboplatin-olaparib followed by olaparib monotherapy versus capecitabine in BRCA1- or BRCA2-mutated HER2-negative advanced breast cancer as first line treatment (REVIVAL): study protocol for a randomized controlled trial. Trials. 2016 Jun 21;17(1):293. doi: 10.1186/s13063-016-1423-0. PMID 27323902